CLINICAL TRIAL: NCT02263261
Title: Reconstructive, Aesthetic and Patient Reported Outcomes Associated With the Use of Flex HD Pliable, Perforated Human Acellular Dermal Matrix in Implant-Based Breast Reconstruction: A Pilot Study
Brief Title: Evaluation of a Human Acellular Dermal Matrix in Post Mastectomy Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTF 13-03
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2015-03

CONDITIONS: Mastectomy; Breast Reconstruction
Keywords: dermal matrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flex HD Pliable Perforated HADM (Other): Single Arm
  Interventions: Other: Flex HD Pliable Perforated HADM

INTERVENTIONS:
Other: Flex HD Pliable Perforated HADM — Human Acellular Dermal Matrix

SUMMARY:
Use of a HADM and implant in post-mastectomy breast reconstruction.

DETAILED DESCRIPTION:
This is a prospective, single-site pilot study in which outcomes associated with the use of Flex HD® Pliable™ Perforated, Human Acellular Dermal Matrix and an implant which are used in post-mastectomy breast reconstruction will be obtained. The data collected will include reconstructive outcomes, aesthetic outcomes and patient-reported outcomes in order to ascertain advantages and disadvantages of using this particular HADM in post-mastectomy breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a single or two-stage, tissue-assisted, implant breast reconstruction
* Mastectomy may be unilateral or bilateral, prophylactic or therapeutic
* Skin incision may be skin sparing, or nipple-areolar sparing
* Have signed written, informed consent
* Be at least 18 years of age

Exclusion Criteria:

* Patients undergoing autologous breast reconstruction
* Patients undergoing breast reconstruction following complications of breast augmentation, mastopexy, breast reduction, or breast conservation surgery (lumpectomy)
* Patients undergoing reconstruction after previously failed attempts at reconstruction
* Patients undergoing autologous breast reconstruction in conjunction with a tissue expander (such as a latissimus dorsi flap, DIEP flap)
* There will be no exclusions based on race or ethnicity
* BMI > 40
* Previous Radiation Treatment. Note: Post-operative radiation treatment does not exclude subjects from study continuation once enrolled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Types and incidence of complications | 6 months post reconstruction
  Documentaiton of any medical and/or surgical problem requiring treatment that arises as a result of the reconstruction procedure

SECONDARY OUTCOMES:
Aesthetic Outcomes | 6 months post reconstruction
  Aesthetic outcomes evaluated by the operating surgeon and two independent board certified plastic surgeons with breast reconstruction expertise
Patient-Reported Outcomes | 6 months post reconstruction
  Use of the Breast Q survey instrument

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Liu Plastic surgery, Mountain View, California
  - Liu Plastic Surgery, San Jose, California